CLINICAL TRIAL: NCT06795113
Title: Optimization of 18F-FDG PET/CT Response Assessment and Prognostic Evaluation Strategies for High-Metabolism Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, GUO RUI, Deputy Chief Physician, Ruijin Hospital
Other Study IDs: RuijinH 2025-1
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma
Keywords: PET/CT; lymphoma; 18F-FDG
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Modeling group, 2000 patients: clinicopathologic feature, post-treatment efficacy, extracted from the electronic medical record system: demographic characteristics (gender, age, ethnicity, family history, etc.), laboratory test results (complete blood count, blood biochemistry), nasopharyngoscopy, pathology, and nuclear medicine examination reports (PET/CT, PET/MR, etc.), tumor characteristics (tumor size, tumor invasion status, lymph node involvement, staging), and treatment plans.
- Validation group, 2000 patients: clinicopathologic feature, post-treatment efficacy, extracted from the electronic medical record system: demographic characteristics (gender, age, ethnicity, family history, etc.), laboratory test results (complete blood count, blood biochemistry), nasopharyngoscopy, pathology, and nuclear medicine examination reports (PET/CT, PET/MR, etc.), tumor characteristics (tumor size, tumor invasion status, lymph node involvement, staging), and treatment plans.

SUMMARY:
To develop a novel method for evaluating treatment response in lymphoma by utilizing PET/CT imaging data from patients with high-metabolic lymphoma. This involves comparing end-of-treatment PET (EOT-PET) with interim PET (iPET) results to establish a new response assessment approach. The aim is to contrast this method with the Lugano classification criteria, providing clinicians with more scientific and accurate tools for response evaluation and prognosis prediction.

DETAILED DESCRIPTION:
This study adopted a multicenter retrospective cohort design. A total of 2,000 patients with highly metabolic lymphoma who underwent PET/CT scans and had clinical data available at Ruijin Hospital, affiliated with Shanghai Jiao Tong University School of Medicine, from June 2013 to December 2023, were selected for model development. The model was validated using an external validation cohort of 2,000 patients with highly metabolic lymphoma who underwent PET/CT scans at other institutions, including West China Hospital of Sichuan University. All patients were required to have undergone 18F-FDG PET/CT scans before treatment, during treatment, and after treatment.

Lesions were manually delineated, and software was used to automatically calculate PET/CT parameters such as SUVmax, metabolic tumor volume (MTV), and total lesion glycolysis (TLG) for primary and metastatic lesions based on 18F-FDG PET/CT. Clinical data for all patients were collected from their medical records, including age, gender, LDH levels, B symptoms, extranodal involvement, IPI score, presence of bulky disease, pathological subtype, and treatment regimen.

Each patient's end-of-treatment PET/CT was compared with baseline PET/CT based on the Lugano criteria to evaluate treatment response, and the results were recorded in Group A. Correspondingly, the end-of-treatment PET/CT was also compared with interim PET/CT to derive a new treatment response evaluation, and the results were recorded in Group B. The treatment response evaluations from Groups A and B were then compared. Statistical analysis was performed to identify patients with inconsistent treatment response evaluations between the two groups. Additionally, it was recorded whether the treatment plan for each patient was altered at the end of first-line therapy based on the treatment response evaluation from Group B.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed high-metabolic lymphoma
2. Underwent 18F-FDG PET/CT imaging before, during, and after treatment
3. Treated with a standard first-line therapeutic regimen according to lymphoma treatment guidelines and individualized patient-specific considerations
4. Complete clinicopathological and follow-up data available Exclusion Criteria

1: History of prior antitumor treatment 2: History of other malignancies 3: Incomplete clinical data or imaging records 4: Presence of other concurrent malignant tumors

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with high-metabolic lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-06-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimization of 18F-FDG PET/CT Response Assessment and Prognostic Evaluation Strategies for High-Metabolism Lymphoma | Before the start of treatment, after 4 cycles of treatment(each cycle is 28 days), and 6-8 weeks after the end of treatment.
  Optimization of 18F-FDG PET/CT Response Assessment and Prognostic Evaluation Strategies for High-Metabolism Lymphoma

SECONDARY OUTCOMES:
Progression-Free Survival | 3 years
  Progression-Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No